# Investigating Patterns in Enrollment and Engagement Among Individuals Coping with Anxiety Disorder: A Study on Anxiety Disorder Clinical Trials

This is an Informed Consent Form For Individuals With Anxiety Disorder in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: November 24, 2023

Informed Consent Form for Participants in an Observational Study

Being invited to complete this form indicates your possible eligibility to participate in an innovative observational clinical study aimed at those suffering from anxiety disorder. This comprehensive guide describes the study's key aims, research methods, and prospective implications, which include both positive and potentially harmful effects. Prior to making a choice, it's critical to fully understand the potential consequences of your engagement, and obtaining advice from your healthcare practitioner can provide vital views. If any component of this material causes you confusion or if you have any questions, please contact the researcher or the appropriate contact person.

Appreciating the Significance of Clinical Trials in Treating Anxiety Disorder

Anxiety disorder is a broad term encompassing a group of mental health conditions characterized by excessive worry, fear, or apprehension that is disruptive to daily life. It's a persistent state of heightened unease, tension, and apprehension that goes beyond normal levels of stress and anxiety.

Clinical trials directed towards anxiety disorder serve a pivotal role in appraising the safety and efficacy of innovative treatments tailored for this condition. They serve as fundamental instruments in assessing whether new therapeutic options surpass existing modalities, providing substantial evidence for their wider adoption.

This study uniquely focuses on understanding the individual experiences of those facing anxiety disorder, actively engaged in a clinical trial integrating medical interventions. The primary objective revolves around a comprehensive examination of trial completion rates and voluntary withdrawals within this specific patient cohort.

## Active Participation in Clinical Trial Surveys

Your active participation is critical in this observational clinical study, in which we encourage you to share your thoughts and experiences. This requires filling out questionnaires every two weeks, which normally take 20-30 minutes of your time. In addition, our team is planning quarterly check-in calls to guarantee continuous support and your continuing participation in the trial.

It is critical to underline that your participation in the survey portion of this experiment is completely optional. You may pick which questions to answer or complete the entire questionnaire based on your choices. Furthermore, you have the option to leave the trial at any moment. Recognizing the personal value of participating in a clinical study, we pledge to give assistance while respecting your privacy.

## Exploring the Significance of Observational Clinical Trials

Participating in this medical trial involves immersion in an observational study, an essential element of clinical research meticulously devised to gather insights through non-intrusive monitoring of patients as they adhere to their treatment protocols.

Researchers will merely observe your experience, thoroughly assessing the outcomes of your condition without altering your treatment plan. This trial structure is crucial for enhancing our comprehension of the inherent progression of a specific medical condition and its effects on individuals experiencing it. Your voluntary engagement in this observational study significantly contributes to advancing medical knowledge and refining care for individuals sharing the same medical condition.

# Setting This Study Apart from Other Clinical Trials for Anxiety Disorder

Acknowledging the distinct nature of this research study is fundamental. It operates purely on an observational basis, indicating that your engagement will not involve

specific therapies or interventions. To make an informed choice about potential participation in a clinical trial, understanding the breadth of anxiety disorder clinical research, including interventional studies encompassing diverse treatment regimens, is pivotal.

Making an informed decision about your potential participation in a clinical trial necessitates an active approach involving thorough research and comparison among trials. Resources such as ClinicalTrials.gov offer comprehensive information about <a href="mailto:anxiety disorder studies">anxiety disorder studies</a>. Furthermore, Power's specialized online platform provides a comprehensive catalog of ongoing <a href="mailto:anxiety disorder clinical trials">anxiety disorder clinical trials</a> actively seeking volunteers. Through meticulous exploration and a comprehensive understanding of various clinical trial categories, you can confidently decide whether or not to participate.

### Securing Your Anonymity in the Research

Protecting the absolute confidentiality of your data remains a core aspect of this study. To ensure your anonymity, please abstain from providing any personal or identifiable information in your questionnaire responses. The committed research team is dedicated to strengthening the privacy and security protocols. Nevertheless, it's important to note that certain legal situations might demand the disclosure of personal data.

# **Prospective Gains**

Participants in this observational clinical research may not immediately perceive benefits, but their involvement could yield considerable long-term impact. The information collected from participants will contribute to formulating future strategies for engaging individuals affected by anxiety disorder, potentially expanding the scope of medical research. Those engaged in this clinical trial have the potential to spark significant advancements in the field of medical research, potentially reshaping the landscape for future anxiety disorder patients.

### Potential Health Effects and Risks

Understanding potential health impacts on participants, particularly in studies assessing new drugs, is essential despite the advancements achieved through clinical trials.

Yet, in observational clinical research, we employ a distinct strategy to mitigate these effects by refraining from administering experimental medications to participants. Our primary focus remains on thorough monitoring and assessing outcomes, ensuring the avoidance of any preventable health risks.

# Reading More About Diversity in Clinical Trials

For those interested in investigating the multifaceted nature of diversity in clinical trials, a plethora of online materials awaits exploration.

Whether your aspiration is to comprehend the intricacies of challenges and opportunities linked to diversity within clinical trials or expand your own perspectives, the following resources can be instrumental in this endeavor:

Hwang, Thomas J., and Otis W. Brawley. "New federal incentives for diversity in clinical trials." *New England Journal of Medicine* 387, no. 15 (2022): 1347-1349.

Corneli, Amy, Emily Hanlen-Rosado, Kevin McKenna, Richardae Araojo, Dawn Corbett, Kaveeta Vasisht, Bernadette Siddiqi, Tesheia Johnson, Luther T. Clark, and Sara B. Calvert. "Enhancing diversity and inclusion in clinical trials." *Clinical Pharmacology & Therapeutics* 113, no. 3 (2023): 489-499.

# Confirmation of Participant

I confirm that I have taken the necessary time to understand and internalize the contents of the informed consent form, whether through independent review or with the assistance of professionals who elucidated its details. I am pleased to state that all my queries have been addressed to my satisfaction.

| Participant Name |
|-----------------------|
| Participant Signature |

| Date |
|---|
| Confirmation of Facilitator |
| I confirm that I conducted an in-depth discussion with the participant, comprehensively elucidating the complexities detailed in this written document. My primary objective was to ensure the participant's thorough understanding of the primary research objectives, the methodology employed, potential risks and benefits, and other essential aspects of the anxiety disorder clinical trial. |
| Printed Name of Assisting Researcher |
| Signature of Assisting Researcher |
| Date |